CLINICAL TRIAL: NCT04573608
Title: The Impact of Minimally Invasive Restorative Techniques on Dental Pain in Pregnant Women: a Randomized Clinical Trial
Brief Title: The Impact of Minimally Invasive Restorative Techniques on Dental Pain in Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Papacarie vs ART in pregnant
Record Dates: First submitted 2020-09-27; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Dental Pain; Patient Satisfaction
Keywords: Minimally Invasive Dentistry
MeSH Terms: conditions — Toothache; Patient Satisfaction | interventions — Papacarie; Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Papacarie-Duo (Experimental)
  Interventions: Drug: Papacarie
- Atraumatic Restorative Treatment (Active Comparator)
  Interventions: Drug: Atraumatic Restorative Treatment

INTERVENTIONS:
Drug: Papacarie — Papacarie was introduced into the cavity using the applicator and left for 40 seconds. A blunt excavator was used to remove the softened dentin. The remaining gel was removed using a cotton pellet. When there was no change in gel color, the cavity was considered caries free. The cavity was then filled with high viscosity glass ionomer cement (GIC) in an encapsulated form (Riva Self-Cure, SDI Limited, Bayswater, VIC, Australia). A mechanical mixer was used to mix the capsule for 10 seconds, the capsule was placed into the applicator to apply the GIC into the cavity. For occluso-proximal cavities, a matrix strip with a wooden wedge was used to provide the appropriate contour of the restoration. A gloved finger was used to apply pressure on the GIC for one minute and occlusion was checked and excess material was removed
  Other Names: Papacarie-Duo
  Arms: Papacarie-Duo
Drug: Atraumatic Restorative Treatment — The tooth was cleaned with a wet cotton pellet to remove debris and plaque. Caries was removed using sharp spoon excavators (Darby-Perry #220/221, #17 DE, Hu-Friedy, Chicago, USA), followed by cleaning the cavity using a small wet cotton pellet and finally dried with a dry cotton pellet. The cavity was considered caries-free when a leather-hard texture was reached and the excavator did not stick anymore. GIC was used to restore the cavity using the same technique described for the other group.
  Other Names: ART
  Arms: Atraumatic Restorative Treatment

SUMMARY:
The aim of the present study was to compare the effectiveness of chemo-mechanical caries removal using Papacarie-Duo and Atraumatic Restorative Treatment (ART) in reducing dental pain in pregnant women.

DETAILED DESCRIPTION:
A randomized controlled clinical trial was conducted in 2019 and included 162 pregnant women visiting family health centers in Alexandria, Egypt with dental pain due to caries not extending to pulp who were randomly assigned into Papacarie-Duo group (n=82) and ART group (n=80) after stratification by number of treated surfaces

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females in the first or second trimester
* Having at least mild dental pain as identified by a score of at least 5mm on a Visual Analogue Scale (VAS) 100-mm-long
* Having at least one carious lesion involving dentine clinically classified as a shallow or medium cavity. This cavity should be accessible to hand instruments (International Caries Detection and Assessment System (ICDAS) score= 5 or 6.

Exclusion Criteria:

* Pregnant women with acute pulpitis, swelling or fistula.
* Uncooperative patients.
* Patients with severe gingivitis (Gingival Index (GI) score=3).
* Patients who are unable to read and/or write and those who refused to participate.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females only
Enrollment: 162 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Pain assessment | up to 6 months
  Difference in pain was measured using Visual Analogue Scale (VAS). The scale is represented by a 100-mm-long horizontal line labeled "no pain" at one end and "worst pain" at the other end. Participants were asked to mark the place on the line representing their level of pain
Satisfaction with treatment | up to 6 months
  Satisfaction with treatment was assessed using two questions: the first question was immediately following treatment: "Was the treatment carried out according to your expectations?" The second question was after 6 months" "Has the treatment solved the problem of your teeth?" Each question was answered on a 10-point scale, with lower values indicating a negative perspective and higher values indicating a positive experience.

SECONDARY OUTCOMES:
Time to remove caries | Procedure (Immediately while treatment)
  Time to remove caries was recorded using a stop watch.

CONTACTS AND LOCATIONS:
Overall Officials: May M Adham, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Mona K ElKashlan, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Wafaa E Abdelaziz, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Family Health Centers, Alexandria, Egypt

REFERENCES:
- [Background] Maru VP, Shakuntala BS, Nagarathna C. Caries Removal by Chemomechanical (Carisolv) vs. Rotary Drill: A Systematic Review. Open Dent J. 2015 Dec 31;9:462-72. doi: 10.2174/1874210601509010462. eCollection 2015. PMID 26962375
- [Background] Gugnani N, Pandit IK, Srivastava N, Gupta M, Sharma M. International Caries Detection and Assessment System (ICDAS): A New Concept. Int J Clin Pediatr Dent. 2011 May-Aug;4(2):93-100. doi: 10.5005/jp-journals-10005-1089. Epub 2010 Apr 15. PMID 27672245
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Derived] Adham MM, El Kashlan MK, Abdelaziz WE, Rashad AS. The impact of minimally invasive restorative techniques on perception of dental pain among pregnant women: a randomized controlled clinical trial. BMC Oral Health. 2021 Feb 18;21(1):76. doi: 10.1186/s12903-021-01432-3. PMID 33602209